CLINICAL TRIAL: NCT06302283
Title: Collateral Effects of Pandemics - Care for Informal Caregivers
Acronym: COLLPAN-3A
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Bonn (Other)
Collaborators: Wuerzburg University Hospital (Other); Johannes Gutenberg University Mainz (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lukas Radbruch, Director Department of Palliative Medicine, University Hospital Bonn, University of Bonn
Other Study IDs: 114/23-EP
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Bereavement
Keywords: Informal Caregiver burden
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family Members or Informal Caregivers: family members or informal caregivers that have cared for a patient with Covid-19 or of a patient who has died in the first phase of the pandemic (March to December 2021)
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey (online or paper) on caregiving burden and bereavement

SUMMARY:
The study is a workpackage in the German research consortium COLLPAN. The study will map collateral effects in terms of psychosocial and spiritual burden of informal caregivers during after the pandemic and identification/mapping of risk factors.It will also map available therapeutic and preventive interventions and relief of this burden for the present situation and for future pandemics.

DETAILED DESCRIPTION:
a scoping literature review will compile evidence on informal caregiver burden during and after the pandemic (PubMed, PsychInfo, Cochrane Database). The aim of the review is to gain knowledge on frequency, severity, source and circumstances of care givers' burden and to identify research and supportive gaps.

The study will recruit family members and care givers of patients with COVID-19 or long-COVID as well as bereaved family members and care givers of patients who have died during the pandemic in order to assess severity of burden. Recruitment will be done in collaboration with the German Association of Undertakers and the Federal Association for Bereavement Care. Family members and caregivers will be asked to complete a survey with instruments on bereavement burden (PG- 13), distress (PHQ-9; GAD-7) and care giver symptoms (IPOS; MIDOS-2). The survey will be available online (using SoSciSurvey platform) or as a paper and pencil version. Survey participants will be invited to in-depth interviews.

Recruitment of 200 participants each for caregiving of COVID-19 patients and bereaved family members will be targeted. Interviews are planned with 30 participants in each group or until saturation is reached.

Based on findings, recommendations on interventions to support family care givers will be developed

ELIGIBILITY:
Inclusion Criteria:

* having cared for a patient with COVID-19 in the first year of the pandemic (March to December 2021)

Exclusion Criteria:

* not fluent in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: family members or caregivers that have cared for patients with COVID-19 or have lost a family member in the first phase of the pandemic (March to December 2021)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bereavement burden | Baseline
  standardized instrument on bereavement burden (PG- 13)
Anxiety | Baseline
  standardized instrument on anxiety (GAD-7)
Depression | Baseline
  standardized instrument on depression (PHQ-9)
Caregiving burden | Baseline
  standardized instrument on caregiver symptoms (MIDOS-2).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Radbruch, MD, Principal Investigator — Department of Palliative Medicine, University Hospital Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No